CLINICAL TRIAL: NCT05405673
Title: A Prospective Cross-sectional Multi-center Study to Assess the Diagnostic Accuracy of a Panel of Bacterial Gene Markers (M3) for Colorectal Advanced Neoplasia
Brief Title: Diagnostic Accuracy of a Panel of Bacterial Gene Markers (M3) for Colorectal Advanced Neoplasia
Acronym: M3-PRO
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other); Aster CMI Hospital (Unknown); Osaka International Cancer Institute (Unknown); Sano hospital (Unknown); Thingangyun Sanpya General Hospital (Unknown); Changi General Hospital (Other); National Taiwan University Hospital (Other); Phramongkutklao College of Medicine and Hospital (Other); St. Mark's Hospital (Unknown); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assistant Professor (clinical), Chinese University of Hong Kong
Other Study IDs: 2022.170
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenoma
Keywords: FIT; Bacterial gene marker; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal neoplasia screening/surveillance cohort: Subjects with average risk of colorectal neoplasias requiring screening/surveillance colonoscopy
  Interventions: Diagnostic Test: Fecal immunochemical test (FIT)

INTERVENTIONS:
Diagnostic Test: Fecal immunochemical test (FIT) — A kind of stool test
  Other Names: Bacterial gene marker test

SUMMARY:
The investigators aim to evaluate and compare the diagnostic accuracy of FIT and the novel panel of bacterial gene markers (Fn, m3, Ch and Bc) collectively named as M3, in detecting colorectal advanced neoplasia.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the one of the most common cancers in Hong Kong with more than 5,500 new cases annually. There is prevailing evidence of increasing trend of young onset CRC globally. Early detection and resection of pre-malignant colorectal neoplasia has shown to reduce CRC-related mortality.

Non-invasive stool tests including guaiac-based faecal occult blood tests (gFOBT) and faecal immunochemical tests (FIT) are the cornerstones of population-based CRC screening programmes. The major limitation of this widely used strategy is its unsatisfactory sensitivities for CRC (79%) and advanced adenomas (AA; 40%). The sensitivity for non-advanced adenomas is even lower than 10%. A large proportion of advanced and non-advanced adenomas will be missed by FIT alone. Therefore, identification of alternative non-invasive test with better sensitivity to detect colorectal neoplasia is warranted.

Multitarget stool DNA test and faecal microbial DNA markers appear to be promising options for CRC screening. Several bacterial gene markers have been identified by metagenome sequencing and reported to be associated with CRC, including Fusobacterium nucleatum (Fn), Clostridium hathewayi (Ch) and Bacteroides clarus (Bc). However, these molecular markers had low accuracy in distinguishing adenomas from normal tissue. Recently, a new Lachnoclostridium gene marker (labelled as 'm3') has been shown to have high diagnostic yield for the detection of colorectal adenomas. In a case-control study of 1012 subjects, a linear increasing trend of m3 level was observed from fecal samples of healthy subjects to those with adenomas and cancers. The overall sensitivity of m3 was significantly higher than FIT in detecting all adenomas (48% vs 9.3%), AA (50.8% vs 16.1%) and non-advanced adenomas (44.2% vs 0%). The diagnostic accuracy of m3 could be further enhanced by combining with a panel of fecal microbial markers composing of Fusobacterium nucleatum (Fn), Bacteroides clarus (Bc), Clostridium hathewayi (Ch) for CRC (82.3%) and adenomas (64.2%). We hypothesized that the combination of these 4 bacterial gene markers (known as M3) is more sensitive than FIT in detecting colorectal advanced neoplasia.

ELIGIBILITY:
Inclusion Criteria:

1. They require elective colonoscopy for colorectal cancer screening or polyp surveillance, or investigation of symptoms (e.g. anemia, change of bowel habit, abdominal pain);
2. Aged ≥18 years old;
3. Written informed consent obtained.

Exclusion Criteria:

1. Contraindications to colonoscopy (e.g. perforation, intestinal obstruction, unstable cardiopulmonary status);
2. Contraindication to polyp resection (e.g. active gastrointestinal bleeding, uninterrupted anticoagulation or dual antiplatelets);
3. Known colorectal cancer or adenoma for staged procedure;
4. Previous colonic resection;
5. Personal history of colorectal cancer;
6. Personal history of polyposis syndrome;
7. Personal history of inflammatory bowel disease;
8. Known pregnancy or lactation;
9. Advanced comorbid conditions (defined as American Society of Anesthesiologists grade 4 or above);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with average risk of colorectal neoplsia requring screening/surveillance colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of bacterial gene markers panel (M3) | 1 month
  The proportion of subjects with true positive results of M3 among those with one of more advanced neoplasia detected in the index colonoscopy.
Sensitivity of FIT/FOBT | 1 month
  The proportion of subjects with true positive results of FIT among those with one of more advanced neoplasia detected in the index colonoscopy.

SECONDARY OUTCOMES:
Sensitivity of M3 for early-stage (stage 1) or invasive (stage 2-4) colorectal cancers | 1 month
  The proportion of subjects with true positive results of M3 among those with early-stage (stage 1) or invasive (stage 2-4) colorectal cancers detected in the index colonoscopy.
Sensitivity of FIT/FOBT for early-stage (stage 1) or invasive (stage 2-4) colorectal cancers | 1 month
  The proportion of subjects with true positive results of FIT among those with early-stage (stage 1) or invasive (stage 2-4) colorectal cancers detected in the index colonoscopy.
Sensitivity of FIT/FOBT for advanced adenomas | 1 month
  The proportion of subjects with true positive results of FIT among those with one or more advanced adenomas detected in the index colonoscopy.
Sensitivity of M3 for advanced adenomas | 1 month
  The proportion of subjects with true positive results of M3 among those with one or more advanced adenomas detected in the index colonoscopy.
Sensitivity of FIT/FOBT for all adenomas | 1 month
  The proportion of subjects with true positive results of FIT among those with all advanced adenomas detected in the index colonoscopy.
Sensitivity of M3 for all adenomas | 1 month
  The proportion of subjects with true positive results of M3 among those with all advanced adenomas detected in the index colonoscopy.
Sensitivity of FIT/FOBT for sessile serrated lesions (SSL) | 1 month
  The proportion of subjects with true positive results of FIT among those with SSLs detected in the index colonoscopy.
Sensitivity of M3 for sessile serrated lesions (SSL) | 1 month
  The proportion of subjects with true positive results of M3 among those with SSLs detected in the index colonoscopy.
Specificity | 1 month
  The proportion of true negative results of M3/FOBT/FIT among those with no adenoma detected in colonoscopy
Positive predictive value (PPV) | 1 month
  The ratio of subjects truly diagnosed as positive to all those who had positive test results
Negative predictive value (NPV) | 1 month
  The ratio of subjects truly diagnosed as negative to all those who had negative test results
Overall diagnostic accuracy | 1 month
  The proportion of correctly classified subjects among all subjects
Microbiota changes in subjects with adenomas or normal findings after polypectomy | 1 month
  Microbiota change measured by qPCR or metagenomic sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No